CLINICAL TRIAL: NCT00082017
Title: Phase II Study of UCN-01 in Relapsed or Refractory Systemic Anaplastic Large Cell and Mature T-Cell Lymphomas
Brief Title: UCN-01 (7-Hydroxystaurosporine) to Treat Relapsed T-Cell Lymphomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IND was withdrawn by CTEP due to low accrual and cost of maintaining the IND.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Wyndham Wilson, M.D., Dr. Wyndham Wilson, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 040173; 04-C-0173; NCT00085319 (obsolete NCT alias)
Record Dates: First submitted 2004-04-28; First posted 2004-04-28 (Estimated); Results first posted 2012-08-29 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Lymphoma, Large-Cell, Ki-1; Lymphoma, T-Cell
Keywords: Protein Kinase Inhibition; Soluble Tac; Gene Expression Profiling; ALK Expression; Apoptosis; Lymphoma; Anaplastic Large Cell Lymphoma; ALCL; T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, T-Cell; Lymphoma | interventions — 7-hydroxystaurosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- UCN-01 for T-cell lymphomas - Cohort 1 - Every 28 days (Experimental): Cycle 1: 45 mg/m^2/day continuous intravenous infusion 1 to 3 days (72 hours) for total dose of 135 mg/m^2
  Cycle 2: 45 mg/m^2/day continuous intravenous infusion 1 to 2 days (36 hours) for total dose of 68 mg/m^2; Repeat cycles every 28 days.
  Interventions: Drug: UCN-01 (7-hydroxystaurosporine)
- UCN-01 for T-cell lymphomas - Cohort 2 -Every 21 days (Experimental): Cycle 1: 45 mg/m^2/day continuous intravenous infusion 1 to 3 days (72 hours) for total dose of 135 mg/m^2
  Cycle 2: 45 mg/m^2/day continuous intravenous infusion 1 to 2 days (36 hours) for total dose of 68 mg/m^2; Repeat cycles every 21 days.
  Interventions: Drug: UCN-01 (7-hydroxystaurosporine)

INTERVENTIONS:
Drug: UCN-01 (7-hydroxystaurosporine) — UCN-01 for relapsed or refractory T-cell lymphomas - Cohort 1, Cycle 1: 45 mg/m^2/day continuous intravenous infusion 1 to 3 days (72 hours) for total dose of 135 mg/m^2 Cycle 2: 45 mg/m^2/day continuous intravenous infusion 1 to 2 days (36 hours) for total dose of 68 mg/m^2; Repeat cycles every 28 days.
  UCN-01 for relapsed or refractory T-cell lymphomas - Cohort 2, Cycle 1: 45 mg/m^2/day continuous intravenous infusion 1 to 3 days (72 hours) for total dose of 135 mg/m^2 Cycle 2: 45 mg/m^2/day continuous intravenous infusion 1 to 2 days (36 hours) for total dose of 68 mg/m^2; Repeat cycles every 21 days.
  Other Names: UCN-01

SUMMARY:
This study will examine the effects of an experimental drug called UCN-01 (7-hydroxystaurosporine) on T-cell lymphomas. UCN-01 inhibits the growth of several different tumor cells, and, in laboratory studies, it has worked particularly well on tumor cells taken from patients with T cell lymphomas.

Patients 9 years of age and older with T cell lymphoma that has relapsed or is not responding to chemotherapy may be eligible for this study. Candidates will be screened with a medical histories and physical examinations, blood and urine tests, electrocardiograms, chest x-rays, and computed tomography (CT) scans of the chest, abdomen and pelvis. Additional tests may be done if clinically indicated, such as positron emission tomography (PET) scans, bone marrow aspirations and biopsies, lumbar punctures (spinal taps) and CT's or magnetic resonance imaging (MRI) scans if there is evidence of central nervous system disease.

Participants are given UCN-01 in 28-day treatment cycles. The drug is given by vein in a continuous 72-hour infusion on the first cycle and in 36-hour infusions on subsequent cycles. The total number of cycles patients receive depends on how well the tumor responds to the drug and how well the patient tolerates drug side effects. Patients who do well may receive treatment for up to 1 year. Patients whose disease worsens with treatment or who do not tolerate the therapy are taken off the study.

Some or all of the screening tests are repeated periodically during the course of treatment to monitor safety and treatment response. X-rays and scans are done every other treatment cycle for the first 6 cycles and then, if the cancer is stable or improving, the interval between these imaging studies is lengthened to every 4 cycles. Patients whose tumors can be safely biopsied undergo this procedure before entering the study and 3 to 5 days after completing the first UCN-01 treatment. Biopsies requiring open surgery (e.g., in the chest or abdomen) are done only if absolutely necessary for medical care. Biopsy tissue, blood, and other fluids are analyzed for gene and protein studies related to lymphoma research.

DETAILED DESCRIPTION:
Background:

* UCN-01 (7-hydroxystaurosporine), a non-specific protein kinase C (PKC) inhibitor appears to have several mechanisms of action including protein kinase C (PKC) isoenzyme inhibition and cyclin dependent kinase activation and inhibition.
* We have demonstrated that cell lines derived from T-cell lymphomas, including those with the t (2; 5) translocation, are very sensitive to UCN-01. The t (2; 5) translocation, associated with three quarters of cases of anaplastic large cell lymphomas (ALCL), is an oncogenic fusion protein - nucleophosmin-anaplastic lymphoma kinase (NPM-ALK).
* Anaplastic lymphoma receptor tyrosine kinase (ALK) is one potential target for UCN-01 action, and anaplastic large cell lymphoma (ALCL) derived SUDHL-1 cells containing the NPM-ALK protein have been shown to be very sensitive to UCN-01.

Objectives:

* To assess the clinical response to UCN-01 and progression-free and overall survival in patients with relapsed or refractory systemic Anaplastic Large Cell and other mature T-cell Lymphomas.
* To assess the effect of UCN-01 on ALK expression in ALCL cells.
* To assess the effect of UCN-01 on soluble tetrameric antibody complexes (TAC) (CD25).
* To evaluate mature T-cell lymphoma malignant cells by complimentary deoxyribonucleic acid (cDNA) microarray.

Eligibility:

* Relapsed or refractory systemic Anaplastic Large Cell Lymphoma (ALCL) with T or Null phenotype or relapsed or refractory mature T-cell lymphomas.
* All patients should have evaluable or measurable disease on entry to study.
* Requires systemic therapy
* Performance Status Eastern Cooperative Oncology Group (ECOG) less than or equal to 2
* Age 7 years or older
* Human immunodeficiency virus (HIV) negative
* Patients should not have received systemic cytotoxic chemotherapy within 3 weeks of study entry.

Design:

* The study will be a Phase II study.
* Patients will receive the first cycle of UCN-01 over 72 hours on days 1-3 and subsequent cycles over 36 hours. Patients with stable disease may receive UCN-01 for up to 1 year beyond achieving maximum response or stable disease, and restaging will be done every 2 cycles for the first 6 cycles and every 4 cycles thereafter.
* Two sequential biopsies will be performed to investigate complimentary deoxyribonucleic acid (cDNA) expression by microarray. Soluble Tac (CD25) will be serially followed in patients.
* For each of the two histologies, this study will be conducted using a Simon two-stage optimal design. Up to 37 patients will be treated.

ELIGIBILITY:
* INCLUSION CRITERIA:

Relapsed or refractory systemic Anaplastic Large Cell Lymphoma (ALCL).

Relapsed or refractory mature T-cell lymphoma to include peripheral T-cell lymphoma unspecified and the following "specified" mature T-cell lymphomas:

Adult T-cell lymphoma; Extranodal natural killer (NK)/T-cell lymphoma,

nasal type; Enteropathy-type T-cell lymphoma;

Hepatosplenic T-cell lymphoma;

Subcutaneous panniculitis-like T-cell lymphoma;

Angioimmunoblastic T-cell lymphoma.

All patients should have evaluable or measurable disease on entry to study.

Histology confirmed by Laboratory of Pathology, National Cancer Institute (NCI).

Performance Status Eastern Cooperative Oncology Group (ECOG) less than or equal to 2.

Age 7 years or older.

Creatinine less than or equal to 1.5 mg/dl or creatinine clearance greater than 50 ml/min for patients at least 18 years.

Pediatric patients should have maximum serum creatinine by age as follows:

* Less than age 7 and less than or equal to age 10 may have a Maximum Serum Creatinine of 1.0 mg/dl
* Less than age10 and less than or equal to age 15 may have a Maximum Serum Creatinine of 1.2 mg/dl
* Age 15 years or older may have a Maximum Serum Creatinine of 1.5 mg/dl

Alternatively, pediatric patients should have a creatinine clearance of greater than 50 m1/min/1.73m^2.

Total bilirubin less than 1.5 x upper limit of normal (ULN) (patients with elevation of total bilirubin consistent with Gilbert's disease are eligible providing they have a normal direct bilirubin);

aspartate aminotransferase (AST) less than or equal to 2.5 x ULN;

absolute neutrophil count (ANC) greater than 500/mm^3;

and platelet greater than or equal to 50,000/mm^3;

unless hematological impairment due to organ involvement by lymphoma.

Provides signed informed consent.

Not pregnant or nursing. This drug has unknown effects in pregnancy and on young infants/children.

Human immunodeficiency virus (HIV) negative.

Willing to use contraception and continue for at least 8 weeks following the last treatment.

No active central nervous system (CNS) lymphoma.

Patients should not have received systemic cytotoxic chemotherapy within 3 weeks of study entry.

Have recovered from the toxic effects of prior therapy to a grade less than or equal to 1.

No history of diabetes mellitus requiring insulin treatment.

No symptomatic pulmonary disease.

No evidence of symptomatic cardiac disease (e.g. symptomatic congestive heart failure, unstable angina pectoris, exertional angina pectoris, cardiac arrhythmia).

Patients may not be concurrently receiving any other investigational agents.

Not a candidate for potentially curative (i.e. transplant) treatment at the time of study entry or the patient has a window of opportunity to receive UCN-01 before a transplant. Patients are required to have considered a transplant. If, having done this, they refuse it, decide against it or decide to wait, they would be eligible for this study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-04-05 (Actual); Primary Completion 2011-09-27 (Actual); Study Completion 2011-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wyndham Wilson, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stein H, Mason DY, Gerdes J, O'Connor N, Wainscoat J, Pallesen G, Gatter K, Falini B, Delsol G, Lemke H, et al. The expression of the Hodgkin's disease associated antigen Ki-1 in reactive and neoplastic lymphoid tissue: evidence that Reed-Sternberg cells and histiocytic malignancies are derived from activated lymphoid cells. Blood. 1985 Oct;66(4):848-58. PMID 3876124
- [Background] Armitage JO, Weisenburger DD. New approach to classifying non-Hodgkin's lymphomas: clinical features of the major histologic subtypes. Non-Hodgkin's Lymphoma Classification Project. J Clin Oncol. 1998 Aug;16(8):2780-95. doi: 10.1200/JCO.1998.16.8.2780. PMID 9704731
- [Background] Falini B, Pileri S, Zinzani PL, Carbone A, Zagonel V, Wolf-Peeters C, Verhoef G, Menestrina F, Todeschini G, Paulli M, Lazzarino M, Giardini R, Aiello A, Foss HD, Araujo I, Fizzotti M, Pelicci PG, Flenghi L, Martelli MF, Santucci A. ALK+ lymphoma: clinico-pathological findings and outcome. Blood. 1999 Apr 15;93(8):2697-706. PMID 10194450
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-C-0173.html

RESULTS

PARTICIPANT FLOW:
Groups:
- UCN-01 for T-cell Lymphomas - Cohort 1-Every 28 Days: Cohort 1 Cycle 1: 45 mg/m^2/day continuous intravenous infusion 1 to 3 days (72 hours) for total dose of 135 mg/m^2
  Cycle 2: 45 mg/m^2/day continuous intravenous infusion 1 to 2 days (36 hours) for total dose of 68 mg/m^2. Repeat cycles every 28 days.
- UCN-01 for T-cell Lymphomas - Cohort 2 Every 21 Days: Cohort 2 Cycle 1: 45 mg/m^2/day continuous intravenous infusion 1 to 3 days (72 hours) for total dose of 135 mg/m^2
  Cycle 2: 45 mg/m^2/day continuous intravenous infusion 1 to 2 days (36 hours) for total dose of 68 mg/m^2; Repeat cycles every 21 days.
Period: Overall Study
Arm/Group | UCN-01 for T-cell Lymphomas - Cohort 1-Every 28 Days | UCN-01 for T-cell Lymphomas - Cohort 2 Every 21 Days
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- UCN-01 for T-cell Lymphomas - Cohort 1&2: Cohort 1 Cycle 1: 45 mg/m^2/day continuous intravenous infusion 1 to 3 days (72 hours) for total dose of 135 mg/m^2
  Cycle 2: 45 mg/m^2/day continuous intravenous infusion 1 to 2 days (36 hours) for total dose of 68 mg/m^2; Repeat cycles every 28 days.
  Cohort 2 Cycle 1: 45 mg/m^2/day continuous intravenous infusion 1 to 3 days (72 hours) for total dose of 135 mg/m^2
  Cycle 2: 45 mg/m^2/day continuous intravenous infusion 1 to 2 days (36 hours) for total dose of 68 mg/m^2; Repeat cycles every 21 days.
Arm/Group | UCN-01 for T-cell Lymphomas - Cohort 1&2
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 14
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.29 (18.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rate
Description: Clinical Response Rate is the percentage of participants with a response assessed by the International Workshop to Standardize Response Criteria. Complete response (CR) is complete disappearance of all detectable clinical and radiographic evidence of disease. Complete response unconfirmed (CRu) is per CR criteria except that if a residual node is >1.5cm, it must have regressed by >75%. Partial response (PR) is no increase in size of nodes, liver or spleen. Progressive disease (PD) is a greater than or equal to 50% increase from nadir. Details re: response criteria, see the protocol link module
Time Frame: 74.5 months
Measure: Number; unit: Percentage of participants
Groups:
- UCN-01 for T-cell Lymphomas - Cohort 1 Every 28 Days: Cycle 1: 45 mg/m^2/day continuous intravenous infusion 1 to 3 days (72 hours) for total dose of 135 mg/m^2 Cycle 2: 45 mg/m^2/day continuous intravenous infusion 1 to 2 days (36 hours) for total dose of 68 mg/m^2. Repeat cycles every 28 days.
- UCN-01 for T-cell Lymphomas - Cohort 2 Every 21 Days: Cycle 1: 45 mg/m^2/day continuous intravenous infusion 1 to 3 days (72 hours) for total dose of 135 mg/m^2 Cycle 2: 45 mg/m^2/day continuous intravenous infusion 1 to 2 days (36 hours) for total dose of 68 mg/m^2; Repeat cycles every 21 days.
Arm/Group | UCN-01 for T-cell Lymphomas - Cohort 1 Every 28 Days | UCN-01 for T-cell Lymphomas - Cohort 2 Every 21 Days
Number analyzed (Participants) | 11 | 9
Percentage of participants
  Complete response | 18 | 0
  Complete response unconfirmed | 0 | 0
  Partial response | 9 | 0
  Progressive disease | 55 | 45
  Stable disease | 9 | 33
  Not evaluable | 9 | 22

2. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time interval from start of treatment to documented evidence of disease progression. Disease progression is assessed by the International Workshop to Standardize Response Criteria for non-Hodgkin's Lymphomas and is defined as a ≥50% increase from nadir in the sum of the products of the greatest diameters of any previously identified abnormal node for partial response's or non-responders or appearance of any new lesion during or at the end of therapy.
Time Frame: 3.6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | UCN-01 for T-cell Lymphomas - Cohort 1 Every 28 Days | UCN-01 for T-cell Lymphomas - Cohort 2 Every 21 Days
Number analyzed (Participants) | 11 | 8
months | 0.8 [0.2 to 2.2] | 0.8 [0.4 to 3.6]

3. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the date of on-study to the date of death from any cause or last follow up.
Time Frame: 55 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | UCN-01 for T-cell Lymphomas - Cohort 1 Every 28 Days | UCN-01 for T-cell Lymphomas - Cohort 2 Every 21 Days
Number analyzed (Participants) | 11 | 8
months | NA [NA to NA] — Confidence interval was not calculated and median was not reached because over half of the participants were alive. | 5.2 [0.7 to 55.0]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 76 months
Measure: Number; unit: Participants
Groups:
- UCN-01 for T-cell Lymphomas - Cohort 1&2: Cohort 1 Cycle 1: 45 mg/m^2/day continuous intravenous infusion 1 to 3 days (72 hours) for total dose of 135 mg/m^2 Cycle 2: 45 mg/m^2/day continuous intravenous infusion 1 to 2 days (36 hours) for total dose of 68 mg/m^2. Repeat cycles every 28 days.
  Cohort 2 Cycle 1: 45 mg/m^2/day continuous intravenous infusion 1 to 3 days (72 hours) for total dose of 135 mg/m^2 Cycle 2: 45 mg/m^2/day continuous intravenous infusion 1 to 2 days (36 hours) for total dose of 68 mg/m^2; Repeat cycles every 21 days.
Arm/Group | UCN-01 for T-cell Lymphomas - Cohort 1&2
Number analyzed (Participants) | 20
Participants | 19

5. Other Pre Specified Outcome: Effect of UCN-01 on Soluble TAC Cluster of Differentiation 25 (CD25)
Description: Soluble TAC (CD25) levels will be assessed in patients with anaplastic large cell lymphoma.
Time Frame: Day 3-5 after drug administration
Population: This outcome measure was not done because data were insufficient to assess for possible effects on soluble TAC (CD25) levels.
Arm/Group | UCN-01 for T-cell Lymphomas - Cohort 1 Every 28 Days | UCN-01 for T-cell Lymphomas - Cohort 2 Every 21 Days
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Evaluation of Mature T-cell Lymphoma Cells by Complementary Double-Stranded Deoxyribonucleic Acid (cDNA) Microarray
Description: Mature T-cells will be analyzed to identify gene expression changes that correlate with loss of a tumor suppressor gene in a human melanoma cell line.
Time Frame: Day 3-5 after drug administration
Population: This outcome measure was not done because there were inadequate samples to evaluate mature T cell lymphoma malignant cells by cDNA microarray.
Arm/Group | UCN-01 for T-cell Lymphomas - Cohort 1 Every 28 Days | UCN-01 for T-cell Lymphomas - Cohort 2 Every 21 Days
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Effect of UCN-01 on Anaplastic Lymphoma Kinase (ALK) Expression in ALCL
Description: Gene expression patterns in participants ALK positive tumors will be assessed.
Time Frame: Day 3-5 after drug administration
Population: This outcome measure was not done because data were insufficient to assess for possible effects of UCN-01 on ALK expression.
Arm/Group | UCN-01 for T-cell Lymphomas - Cohort 1 Every 28 Days | UCN-01 for T-cell Lymphomas - Cohort 2 Every 21 Days
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 77 months
Arm/Group | UCN-01 for T-cell Lymphomas - Cohort 1&2
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 19/20
Other Adverse Events (participants affected / at risk) | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UCN-01 for T-cell Lymphomas - Cohort 1&2 (N=20)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 6 (9)
Alkaline phosphatase increased (Investigations) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 11 (21)
Anorexia (Metabolism and nutrition disorders) | 4 (5)
Anxiety (Psychiatric disorders) | 1 (1)
Arteritis infective (Infections and infestations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 9 (12)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 8 (8)
Cardiac disorders-Other, specify (Cardiac disorders) | 2 (2) — 1. troponin-due to pericarditis 2. murmur
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
CPK increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 7 (8)
Fever (General disorders) | 3 (3)
Headache (Nervous system disorders) | 7 (12)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (22)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (6)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (5)
Hypotension (Vascular disorders) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Infection with normal absolute neutrophil count (ANC) or grade 1 or 2 neutrophils: Blood
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (14)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (10)
Neutrophil count decreased (Investigations) | 6 (12)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Platelet count decreased (Investigations) | 8 (9)
Proteinuria (Renal and urinary disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Renal and urinary disorders - Other, specify (dysuria) (Renal and urinary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Serum amylase increased (Investigations) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 3 (4)
Small intestine infection (Infections and infestations) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (18)
Weight loss (Investigations) | 1 (3)
White blood cell decreased (Investigations) | 8 (13)
Death (hypercalcemia) (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UCN-01 for T-cell Lymphomas - Cohort 1&2 (N=20)
abdominal pain (Gastrointestinal disorders) | 4 (5)
Activated partial thromboplastin time prolonged (Investigations) | 3 (6)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (6)
Alkaline phosphatase increased (Investigations) | 3 (3)
Allergic rhinitis (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (6)
Bruising (Injury, poisoning and procedural complications) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 5 (7)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine increased (Investigations) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ear and labyrinth disorders-Other, specify (fullness-R ear) (Ear and labyrinth disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Edema trunk (General disorders) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
GGT increased (Investigations) | 2 (3)
Headache (Nervous system disorders) | 2 (3)
Hepatobiliary disorders-Other, specify (hyperbilirubinemia) (Hepatobiliary disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hypermagnesemia (Investigations) | 4 (4)
Hypertension (Vascular disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (12)
Hypokalemia (Metabolism and nutrition disorders) | 6 (11)
Hypomagnesemia (Metabolism and nutrition disorders) | 8 (13)
Hyponatremia (Metabolism and nutrition disorders) | 9 (20)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (12)
Hypotension (Vascular disorders) | 5 (6)
Hypothermia (General disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infections and infestations - Other (Infection with normal ANC or grade 1 or 2 neutrophils: Blood) (Infections and infestations) | 4 (4) — Infection with grade 3 or 4 neutrophils (ANC) < 1.0 x 10e9/L): skin (cellulitis), Infection with normal ANC or grade 1 or 2 neutrophils: peritoneal cavity, Infection with grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Lung (pneumonia)
Injection site reaction (General disorders) | 1 (2)
INR increased (Investigations) | 1 (1)
Investigations-Other, specify (Investigations) | 1 (2)
Lymphocyte count decreased (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (2)
Platelet count decreased (Investigations) | 3 (5)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Seizure (Nervous system disorders) | 1 (1)
Serum amylase increased (Investigations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (4)
Skin and subcutaneous tissue disorders-Other, specify (hives) (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (3)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (7)
White blood cell decreased (Investigations) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No